CLINICAL TRIAL: NCT03283397
Title: A Phase IIIb, Multi-center, International, Randomized, Assessor-blind, Active-controlled Parallel Arm Clinical Study to Evaluate the Efficacy, Safety and Tolerability of Neuropeptide Combination of Metenkefalin and Tridecactide (EK-12) in Comparison to Interferon Beta-1a (REBIF®) in Patients With Relapsing Remitting Multiple Sclerosis (RRMS)
Brief Title: A Phase IIIb, Multicenter, International Study to Evaluate the Efficacy, Safety and Tolerability of EK-12 in Patients With RRMS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: During the Covid-19 pandemic, the study was unable to enrol further patients.
Sponsor: Bosnalijek D.D (Industry)
Collaborators: MonitorCRO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RAP-CS-01
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2023-02

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to one of the two treatment arms and will be observed during the treatment period of 144 weeks
Who Masked: Outcomes Assessor
Masking Description: A blinded examining neurologist/assessor will conduct neurological examinations, relapse and EDSS evaluations at each site. Treating investigators will not be blinded to the study treatment. Additionally, blinded evaluation of MRI scans will be performed at a central reading facility in which, anonymized and standardized images of patient with RRMS will be read by a treatment blinded assessor and data will be implemented in a post-hoc analysis for selected time-points.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EK-12 (Experimental): This arm will be treated with 12 mg EK-12 in 2 mL 0.9 % NaCl solution (SC, three times per week) for 144 weeks
  Interventions: Drug: EK-12
- INF Beta-1a (Active Comparator): This arm will be treated with 44 mg INF Beta-1a in 0.5 mL solution (SC, three times per week) for 144 weeks
  Interventions: Drug: INF beta-1a

INTERVENTIONS:
Drug: EK-12 — 10 mg metenkefalin acetate + 2 mg tridecactide acetate in 2 mL 0.9 % NaCl solution.
  Arms: EK-12
Drug: INF beta-1a — Active substance is INF beta-1a, 44 mcg in 0.5 mL solution
  Arms: INF Beta-1a

SUMMARY:
Multiple sclerosis is a chronic autoimmune, inflammatory neurological disease of the central nervous system. It is the most common disabling neurologic disease of young people. This study is planned for the evaluation of efficacy, safety and tolerability of neuropeptide combination of metenkefalin and tridecactide (EK-12) as compared to INF beta-1a (REBIF®) in patients with RRMS. The primary objective of this study is to prove the superiority of efficacy of neuropeptide combination of metenkefalin and tridecactide (EK-12) compared to INF beta-1a (REBIF®) in patients with RRMS on the basis of annualized protocol defined relapse rate by 144 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients from both genders with a confirmed and documented diagnosis of MS as defined by the Revised McDonald criteria (2010), with relapse onset disease or a relapsing-remitting disease course, between 18 and 55 years of age at screening (inclusive).
2. Ambulatory patients with EDSS score of 0 to 4.5 at both screening and randomization visits.
3. Patients who meet one of the following disease activity criteria:

   * At least 1 documented relapse within the last 12 months prior to screening or;
   * At least 1 documented relapse occurred within the last 24 months prior to screening and documented evidence of at least 1 Gadolinium Enhancing (GdE) lesion on brain MRI scan within the last 12 months prior to randomization.
4. Patients with a confirmed stable neurological condition, who are relapse-free and not on a corticosteroid treatment [intravenous (IV), intramuscular (IM) and/or per os (PO)] or adrenocorticotrophic hormone (ACTH) treatment, at least 30 days prior to randomization.
5. Women of child-bearing potential (e.g. women who are not postmenopausal or surgically sterilized) must practice an acceptable method of birth control for 30 days before taking the study drug and two acceptable methods of birth control during the duration of the study and until 30 days after the last dose of study medication. Acceptable methods of birth control include: intrauterine devices, barrier method (condom with spermicide or diaphragm with spermicide) and hormonal methods of birth control (e.g. oral contraceptive, contraceptive patch, and long-acting injectable contraceptive).
6. Patients must be able to sign and date a written Informed Consent Form (ICF) prior to entering the study.
7. Patients must be willing and able to comply with the study protocol requirements for the duration of the study

Exclusion Criteria:

1. Patients with progressive forms of MS.
2. Patients with disease duration of ≥10 years.
3. Inability to complete an MRI examination. Contraindications for MRI examination include but are not restricted to overweight, pacemaker, cochlear implants, presence of foreign substances in the eye, intracranial vascular clips, surgery within 6 weeks of entry into the study, coronary stent implanted within 8 weeks prior to the time of the intended MRI, etc.
4. Patients with neuromyelitis optica (NMO) or NMO spectrum disorders.
5. Use of experimental or investigational drugs and/or participation in drug clinical studies within 6 months prior to randomization.
6. Use of immunosuppressive agents or cytotoxic agents, including cyclophosphamide within 6 months prior to randomization.
7. Use of either of the following agents within 2 years prior to randomization: natalizumab, rituximab, ocrelizumab, atacicept, belimumab, or ofatumumab.
8. Use of teriflunomide within 2 years prior to randomization, except if active washout (with either cholestyramine or activated charcoal) was done 2 months or more prior to randomization.
9. Previous treatment with glatiramer acetate, interferon-beta (either 1a or 1b), fingolimod, dimethyl fumarate or intravenous immunoglobulin (IVIG) within 2 months prior to randomization.
10. Chronic (more than 30 consecutive days) systemic (IV, IM or PO) corticosteroid treatment within 30 days prior to randomization.
11. Previous use of mitoxantrone, cladribine, or alemtuzumab.
12. Previous use of EK-12.
13. Previous total body irradiation or total lymphoid irradiation.
14. Previous stem cell treatment, autologous bone marrow transplantation or allogeneic bone marrow transplantation.
15. Use of moderate/strong inhibitors of CYP3A4 within 2 weeks prior to randomization (Appendix VII provides a list of such medications that are disallowed prior to and during the study).
16. Use of inducers of CYP3A4 within 2 weeks prior to randomization (Appendix VII provides a list of such medications that are disallowed prior to and during the study).
17. Pregnancy or breastfeeding.
18. Serum levels ≥3x upper limit of the normal range (ULN) of either alanine aminotransferase (ALT) or aspartate aminotransferase (AST) at screening.
19. Serum direct bilirubin ≥2x ULN at screening.
20. Patients with clinically significant or unstable medical or surgical condition or any other condition that cannot be well controlled by the allowed medications permitted by the study protocol that would preclude safe and complete study participation, as determined by medical history, physical examinations, Electrocardiography (ECG), laboratory tests, MRI scan or chest X-ray. Such conditions may include:

    1. A major cardiovascular event (e.g. myocardial infarction, acute coronary syndrome, de-compensated congestive heart failure, pulmonary embolism, coronary revascularization) that occurred during the past 6 months prior to randomization.
    2. Any acute pulmonary disorder
    3. A Central Nervous System (CNS) disorder other than MS that may jeopardize the patient's participation in the study, including such disorders that are demonstrated at the baseline MRI scan.
21. Chronic renal insufficiency as Glomerular Filtration Rate (GFR) ≤60 mL/min at the screening visit.
22. Patients who use haloperidol or dopamine antagonists.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 301 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Superiority of efficacy of EK-12 to interferon beta-1a in patients with RRMS | weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144
  The primary objective of this study is to prove the superiority of efficacy of neuropeptide combination of metenkefalin and tridecactide (EK-12) compared to interferon beta-1a (INF beta-1a, 44 mcg, REBIF®) in patients with RRMS on the basis of annualized protocol defined relapse rate (ARR) by 144 weeks.

SECONDARY OUTCOMES:
EDSS score | weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144
  slowing the progression of disability, assessed by EDSS score
clinical attacks | weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144
  reducing the rate of clinical attacks
T2 lesions | weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144
  reducing the total number of new and/or enlarging T2-hyperintense lesions
T1 lesions | weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144
  reducing the total number of Gd (+) T1 lesions on MRI scan

CONTACTS AND LOCATIONS:
Overall Officials: Husnu Efendi, Prof, Principal Investigator — Kocaeli University
Locations (1):
- Kocaeli University, Faculty of Medicine, Department of Neurology, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No